CLINICAL TRIAL: NCT03473925
Title: A Phase II Study of Navarixin (MK-7123) in Combination With Pembrolizumab (MK-3475) in Participants With Selected Advanced/Metastatic Solid Tumors
Brief Title: Efficacy and Safety Study of Navarixin (MK-7123) in Combination With Pembrolizumab (MK-3475) in Adults With Selected Advanced/Metastatic Solid Tumors (MK-7123-034)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7123-034; MK-7123-034 (Other: Merck Protocol Number)
Record Dates: First submitted 2018-03-08; First posted 2018-03-22 (Actual); Results first posted 2022-06-29 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-07

CONDITIONS: Solid Tumors; Non-small Cell Lung Cancer; Castration Resistant Prostate Cancer; Microsatellite Stable Colorectal Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — navarixin; 2-hydroxy-N,N-dimethyl-3-(2-((1-(5-methylfuran-2-yl)propyl)amino)-3,4-dioxocyclobut-1-enylamino)benzamide; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Navarixin 30 mg + Pembrolizumab 200 mg (Experimental): Participants received 30 mg navarixin via oral capsules once daily, plus 200 mg pembrolizumab via IV infusion on Day 1 of each 3-week cycle for up to 35 administrations (up to approximately 2 years
  Interventions: Drug: Navarixin; Biological: Pembrolizumab
- Navarixin 100 mg + Pembrolizumab 200 mg (Experimental): Participants received 100 mg navarixin via oral capsules once daily, plus 200 mg pembrolizumab via IV infusion on Day 1 of each 3-week cycle for up to 35 administrations (up to approximately 2 years).
  Interventions: Drug: Navarixin; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Navarixin — Oral capsules
  Other Names: MK-7123; SCH 527123
Biological: Pembrolizumab — Intravenous infusion
  Other Names: MK-3475

SUMMARY:
The purpose of this study is to assess the efficacy and safety of navarixin (MK-7123) in combination with pembrolizumab (MK-3475) in adults with one of three types of solid tumors: Programmed Death-Ligand 1 (PD-L1) positive refractory non-small cell lung cancer (NSCLC), castration resistant prostate cancer (CRPC) or microsatellite stable (MSS) colorectal cancer (CRC).

ELIGIBILITY:
Inclusion Criteria:

All Participants

* Has one of the following histologically- or cytologically-confirmed advanced/metastatic solid tumors: NSCLC, CRPC, or MSS CRC, by pathology report and has received, or been intolerant to, or has been ineligible for all treatment known to confer clinical benefit.
* Has Stage III or Stage IV disease that is not surgically resectable.
* Has measurable disease by RECIST 1.1 criteria as assessed by the local site investigator/radiology.
* Has supplied tumor tissue from either a newly obtained biopsy or an archival specimen for biomarker analysis.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Male participants must agree to use contraception during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.
* Female participants must agree to follow the contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment.
* Demonstrates adequate organ function.

Non-small Cell Lung Cancer (NSCLC) Participants

* Has histologically or cytologically confirmed diagnosis of Stage IV metastatic NSCLC.
* Has progressed on treatment with an anti-Programmed Death-Ligand 1 (PD-L1) monoclonal antibody (mAb) administered either as monotherapy, or in combination with other checkpoint inhibitors or other therapies. PD-L1 treatment progression is defined by meeting all of the following criteria: a) Has received ≥2 doses of an approved anti-PD-L1 mAb; b) Has demonstrated disease progression after anti-PD-L1 as defined by RECIST 1.1; c) Progressive disease has been documented within 12 weeks from the last dose of anti-PD-L1 mAb.

Castration Resistant Prostate Cancer (CRPC) Participants

* Has histologically- or cytologically-confirmed adenocarcinoma of the prostate. Components of small cell prostate cancer are permitted.
* Has prostate cancer progression on the most recent treatment, as determined by the investigator, by means of one of the following: a) Prostate-Specific Antigen (PSA) progression using local laboratory values as defined by a minimum of 2 rising PSA levels with an interval of ≥1 week between each assessment where the PSA value at screening should be ≥2 ng/mL; b) Radiographic disease progression in soft tissue based on RECIST 1.1 criteria with or without PSA progression; c) Radiographic disease progression in bone defined as the appearance of 2 or more new bone lesions on bone scan with or without PSA progression.
* Has progressed on at least one second generation anti-androgen therapy (e.g., enzalutamide, abiraterone).
* Has ongoing androgen deprivation with serum testosterone <50 ng/dL (<2.0 nM).

Microsatellite Stable Colorectal Cancer (MSS-CRC) Participants

* Has a histologically proven locally advanced unresectable or metastatic (Stage IV) CRC.
* Has locally confirmed (MSS) CRC; participants with microsatellite instability-high (MSI-H) or microsatellite unstable CRC are not eligible.
* Has been previously treated with standard therapies, which must include fluoropyrimidine, oxaliplatin, and irinotecan.

Exclusion Criteria:

* Has a known additional malignancy that is progressing or has required active treatment within the past 2 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging, clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
* Has had a severe hypersensitivity reaction to treatment with any mAb or components of the study treatment(s).
* Has an active autoimmune disease that has required systemic treatment in the past 2 years except vitiligo or resolved childhood asthma/atopy. Participants who have previously been permanently discontinued from PD-(L)1 therapy due to immune related side effects are not eligible for this study.
* Has an active infection requiring systemic therapy.
* Has symptomatic ascites or pleural effusion.
* Has interstitial lung disease that required oral or intravenous glucocorticoids to assist with management.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has undergone prior allogeneic hematopoietic stem cell transplantation within the last 5 years. Note: Participants who have had a stem cell transplant >5 years ago are eligible as long as there are no symptoms of graft-versus-host disease (GVHD).
* Has a known history of human immunodeficiency virus (HIV) infection.
* Has a known history of Hepatitis B or known active Hepatitis C virus infection.
* Has a history or current evidence of a gastrointestinal condition (e.g. inflammatory bowel disease, Crohn's disease, ulcerative colitis) or impaired liver function or diseases that in the opinion of the Investigator may significantly alter the absorption or metabolism of oral medications; any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, make administration of the study drugs hazardous, or make it difficult to monitor AEs such that it is not in the best interest of the participant to participate, in the opinion of the treating Investigator.
* Is pregnant or expecting to conceive or father children within the projected duration of the study.
* Has undergone major surgery and has not recovered adequately from any toxicity and/or complications from the intervention prior to starting study treatment.
* Has CRPC or MSS CRC and has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has been treated with an agent directed to another stimulatory or co-inhibitory Tcell receptor (e.g. cytotoxic T-lymphocyte protein 4 [CTLA-4], tumor necrosis factor receptor superfamily, member 4 [OX 40], tumor necrosis factor receptor superfamily member 9 [CD137]).
* Has received prior systemic anti-cancer therapy including investigational agents or has used an investigational device within 28 days prior to the first dose of study treatment.
* Has received prior radiotherapy (not to target lesions) within 2 weeks of start of study treatment.
* Is expected to require any other form of antineoplastic therapy while on study.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy in excess of replacement doses (prednisone ≤10 mg/day is acceptable), or on any other form of immunosuppressive medication.
* Has received a live-virus vaccine within 30 days prior to first dose of study treatment.
* Has been previously treated with a chemokine receptor 2 (CXCR2) inhibitor (e.g. AZD5069, reparixin, danirixin, LY3041658 Ab, HuMax-IL8, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (14):
- United States (5):
  - Honor Health ( Site 0005), Scottsdale, Arizona
  - Florida Cancer Specialists ( Site 0003), Sarasota, Florida
  - University of Maryland ( Site 0008), Baltimore, Maryland
  - Henry Ford Health System ( Site 0006), Detroit, Michigan
  - Duke University Medical Center ( Site 0004), Durham, North Carolina
- Australia (3):
  - Blacktown Hospital Western Sydney Local Health District ( Site 0024), Blacktown, New South Wales
  - Scientia Clinical Research ( Site 0021), Randwick, New South Wales
  - Peter MacCallum Cancer Centre ( Site 0023), Melbourne, Victoria
- Canada (2):
  - Princess Margaret Cancer Centre ( Site 0031), Toronto, Ontario
  - Jewish General Hospital ( Site 0032), Montreal, Quebec
- Sourasky Medical Center ( Site 0012), Tel Aviv, Israel
- South Korea (3):
  - Seoul National University Bundang Hospital ( Site 0043), Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital ( Site 0042), Seoul
  - Severance Hospital Yonsei University Health System ( Site 0041), Seoul

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Armstrong AJ, Geva R, Chung HC, Lemech C, Miller WH Jr, Hansen AR, Lee JS, Tsai F, Solomon BJ, Kim TM, Rolfo C, Giranda V, Ren Y, Liu F, Kandala B, Freshwater T, Wang JS. CXCR2 antagonist navarixin in combination with pembrolizumab in select advanced solid tumors: a phase 2 randomized trial. Invest New Drugs. 2024 Feb;42(1):145-159. doi: 10.1007/s10637-023-01410-2. Epub 2024 Feb 7. PMID 38324085

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults with one of the following types of solid tumors: Programmed Death-Ligand 1 (PD-L1) positive refractory non-small cell lung cancer (NSCLC), castration resistant prostate cancer (CRPC) or microsatellite stable (MSS) colorectal cancer (CRC), were enrolled in this study.
Groups:
- Navarixin 30 mg + Pembrolizumab 200 mg: Participants received 30 mg navarixin via oral capsules once daily, plus 200 mg pembrolizumab via intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 administrations (up to approximately 2 years).
Period: Overall Study
Arm/Group | Navarixin 30 mg + Pembrolizumab 200 mg | Navarixin 100 mg + Pembrolizumab 200 mg
Started (Randomized) | 52 | 55
Treated | 51 | 54
Completed | 0 | 0
Not Completed | 52 | 55
Not completed — Death | 48 | 44
Not completed — Sponsor Decision | 2 | 7
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Not Treated | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Navarixin 30 mg + Pembrolizumab 200 mg: Participants received 30 mg navarixin via oral capsules once daily, plus 200 mg pembrolizumab via IV infusion on Day 1 of each 3-week cycle for up to 35 administrations (up to approximately 2 years).
- Total: Total of all reporting groups
Arm/Group | Navarixin 30 mg + Pembrolizumab 200 mg | Navarixin 100 mg + Pembrolizumab 200 mg | Total
Number analyzed (Participants) | 51 | 54 | 105
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.1 (13.3) | 62.8 (13.0) | 63.4 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 37 | 41 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 49 | 54 | 103
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 14 | 11 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 36 | 39 | 75
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: ORR is defined as the percentage of participants who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. ORR was estimated using an exact method based on the binomial distribution, and the 95% confidence interval was estimated by the method of Clopper-Pearson.
Time Frame: Up to approximately 2 years
Population: All participants with a baseline scan that demonstrated measurable disease by the investigator's assessment, and who were administered at least 1 dose of study medicine.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Navarixin 30 mg + Pembrolizumab 200 mg | Navarixin 100 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 51 | 54
Percentage of participants | 3.9 [0.5 to 13.5] | 1.9 [0.0 to 9.9]

2. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs) During Treatment Cycle 1
Description: The following toxicities are considered a DLT, assessed as related to study treatment: Grade 4 non-hematologic toxicity, Grade 4 anemia, Grade 3 anemia lasting >7 days or requiring transfusion, Grade 4 hematologic toxicity lasting ≥7 days, except thrombocytopenia, a) Grade 4 thrombocytopenia of any duration, b) Grade 3 thrombocytopenia associated with bleeding, Grade 3 non-hematologic toxicity lasting >3 days, any Grade 3 or Grade 4 non-hematologic laboratory value if: medical intervention is required or the abnormality leads to hospitalization or persists for >72 hours, Liver test abnormalities: Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3X Upper Limit of Normal (ULN) with total bilirubin (TBL) >2X ULN with no elevation in alkaline phosphatase (AP <2X ULN), Grade 3 or Grade 4 febrile neutropenia, inability to administer ≥75% of the planned navarixin dose due to drug-related tolerability, delay in Cycle 2 start by >2 weeks due to toxicity
Time Frame: Up to 21 days
Population: Participants who complete cycle 1 without any discontinuation, or discontinues from the study prior to completing all the safety evaluations in cycle 1 due to treatment-related adverse events, or if participants receive >=75% of the total pembrolizumab infusion and/or navarixin in cycle, or If the participants experience any DLT in AE.
Measure: Count of Participants; unit: Participants
Arm/Group | Navarixin 30 mg + Pembrolizumab 200 mg | Navarixin 100 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 48 | 48
Participants | 2 | 3

3. Primary Outcome: Number of Participants Who Experience at Least One Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment.
Time Frame: Up to approximately 27 months
Population: All participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Navarixin 30 mg + Pembrolizumab 200 mg | Navarixin 100 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 51 | 54
Participants | 50 | 54

4. Primary Outcome: Number of Participants Who Discontinue Study Treatment Due to an AE
Description: as for outcome 3
Time Frame: Up to approximately 2 years
Population: All participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Navarixin 30 mg + Pembrolizumab 200 mg | Navarixin 100 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 51 | 54
Participants | 4 | 6

5. Secondary Outcome: Objective Response Rate (ORR) Per Modified RECIST 1.1 for Immune-based Therapeutics (iRECIST)
Description: An objective response is defined as an immune-based Complete Response (iCR: Disappearance of all target lesions) or immune-based Partial Response (iPR: At least a 30% decrease in the sum of diameters of target lesions). ORR will be assessed by the investigator based on iRECIST following administration of navarixin in combination with pembrolizumab. The percentage of participants with progressive disease per RECIST 1.1 who experience an iCR or iPR are presented.
Time Frame: Up to approximately 2 years
Population: All participants with a baseline scan that demonstrated measurable disease by the investigator's assessment, and who were administered at least 1 dose of study medicine. Only participants with progressive disease per RECIST 1.1 are included.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Navarixin 30 mg + Pembrolizumab 200 mg | Navarixin 100 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 43 | 41
Percentage of participants
  iComplete Response (iCR) | 0.0 [0.0 to 8.2] | 0.0 [0.0 to 8.6]
  iPartial Response (iPR) | 0.0 [0.0 to 8.2] | 0.0 [0.0 to 8.6]

6. Secondary Outcome: Progression-free Survival (PFS) Per RECIST 1.1
Description: PFS is defined as the time from the first dose of study treatment to the first confirmed documented disease progression, or death due to any cause, whichever occurs first. Per RECIST 1.1, progressive disease is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions is also considered progression. Median PFS per RECIST 1.1 was assessed by the investigator from product-limit (Kaplan-Meier) method for censored data in participants with microsatellite stable colorectal cancer (CRC); with castration-resistant prostate cancer (CRPC), and with programmed cell death ligand 1 (PD-[L]1) refractory non-small cell lung cancer (NSCLC).
Time Frame: Up to approximately 2 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Navarixin 30 mg + Pembrolizumab 200 mg | Navarixin 100 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 51 | 54
Months
  CRC: number analyzed (Participants) | 19 | 21
  CRC | 1.8 [1.0 to 2.0] | 1.9 [1.6 to 2.0]
  CRPC: number analyzed (Participants) | 20 | 20
  CRPC | 2.1 [1.9 to 4.1] | 2.1 [1.9 to 4.5]
  NSCLC: number analyzed (Participants) | 12 | 13
  NSCLC | 2.4 [1.6 to 10.2] | 2.1 [1.9 to 2.4]

7. Secondary Outcome: PFS Per iRECIST
Description: PFS is defined as the time from the first dose of study treatment to the first documented disease progression or death due to any cause, whichever occurs first. Per iRECIST, progressive disease (PD) is defined as ≥20% increase in the sum of diameters of target lesions. Disease progression is to be confirmed by a consecutive assessment at least 4-8 weeks after first documentation and will be assessed by the investigator. Median PFS per iRECIST was assessed by the investigator from product-limit (Kaplan-Meier) method for censored data in participants with microsatellite stable colorectal cancer (CRC); with castration-resistant prostate cancer (CRPC), and with programmed cell death ligand 1 (PD-[L]1) refractory non-small cell lung cancer (NSCLC).
Time Frame: Up to approximately 2 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Navarixin 30 mg + Pembrolizumab 200 mg | Navarixin 100 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 51 | 54
Months
  CRC: number analyzed (Participants) | 19 | 21
  CRC | 4.1 [2.1 to 7.1] | 6.2 [3.3 to 14.4]
  CRPC: number analyzed (Participants) | 20 | 20
  CRPC | 7.9 [5.0 to 8.6] | 5.2 [3.0 to 11.5]
  NSCLC: number analyzed (Participants) | 12 | 13
  NSCLC | 11.9 [3.2 to 17.5] | 7.0 [2.4 to 14.4]

8. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the first dose of study treatment to death due to any cause. Median OS was assessed from product-limit (Kaplan-Meier) method for censored data in participants with microsatellite stable colorectal cancer (CRC); with castration-resistant prostate cancer (CRPC), and with programmed cell death ligand 1 (PD-[L]1) refractory non-small cell lung cancer (NSCLC).
Time Frame: Up to approximately 2 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Navarixin 30 mg + Pembrolizumab 200 mg | Navarixin 100 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 51 | 54
Months
  CRC: number analyzed (Participants) | 19 | 21
  CRC | 6.5 [3.0 to 9.7] | 8.0 [5.7 to 14.4]
  CRPC: number analyzed (Participants) | 20 | 20
  CRPC | 10.8 [7.9 to 13.4] | 11.2 [3.7 to 23.0]
  MSCLC: number analyzed (Participants) | 12 | 13
  MSCLC | 13.0 [3.2 to 18.0] | 12.0 [2.4 to 19.9]

9. Secondary Outcome: Absolute Neutrophil Counts (ANC)
Description: Peripheral blood neutrophil counts were performed at Cycle 1 Day 3: Predose, to determine the concentration of ANC.
Time Frame: Day 3: Predose
Population: Participants who complied with the protocol sufficiently to ensure that their data will be likely to exhibit the effects of treatment, according to the underlying scientific model. Compliance includes such considerations as exposure to treatment, availability of measurements, and the absence of major protocol violations
Measure: Mean (95% Confidence Interval); unit: 10^9 cells/L
Arm/Group | Navarixin 30 mg + Pembrolizumab 200 mg | Navarixin 100 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 50 | 51
10^9 cells/L | 3.6 [3.03 to 4.12] | 3.2 [2.50 to 3.84]

10. Secondary Outcome: Navarixin Area Under the Plasma Concentration-Time Curve (AUC) From Time 0 to Infinity (AUC0-inf)
Description: Plasma samples from participants with selected advanced/metastatic solid tumors were collected to determine the navarixin plasma AUC0-inf
Time Frame: Cycle 1 Day 1: Predose & 1, 2, 4, 6 & 8-12 hours postdose; Cycle 1 Days 3 & 8: Predose & 6-12 hours postdose; Cycle 2 Day 1: Predose & 1, 2, 4, 6 & 8-12 hours postdose (Up to approximately 23 days)
Population: Participants with available AUC-inf data, who complied with the protocol sufficiently to ensure that their data was likely to exhibit the effects of treatment, according to the underlying scientific model. Compliance includes, but is not limited to, exposure to treatment, availability of measurements, and absence of major protocol violations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Navarixin 30 mg + Pembrolizumab 200 mg | Navarixin 100 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 38 | 27
h*ng/mL | 523 (39.5) | 1200 (47.5)

11. Secondary Outcome: Navarixin Area Under the Plasma Concentration-Time Curve From Time 0 to Last (AUC0-last)
Description: Plasma samples from participants with selected advanced/metastatic solid tumors were collected to determine the navarixin plasma AUC0-last.
Time Frame: Cycle 1 Day 1: Predose & 1, 2, 4, 6 & 8-12 hours postdose; Cycle 1 Days 3 & 8: Predose & 6-12 hours postdose; Cycle 2 Day 1: Predose & 1, 2, 4, 6 & 8-12 hours postdose(Up to approximately 23 days)
Population: Participants with available AUC-last data, who complied with the protocol sufficiently to ensure that their data was likely to exhibit the effects of treatment, according to the underlying scientific model. Compliance includes, but is not limited to, exposure to treatment, availability of measurements, and absence of major protocol violations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Navarixin 30 mg + Pembrolizumab 200 mg | Navarixin 100 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 45 | 46
h*ng/mL | 451 (35.7) | 961 (45.9)

12. Secondary Outcome: Navarixin Maximum Plasma Concentration (Cmax)
Description: Plasma samples from participants with selected advanced/metastatic solid tumors were collected to determine the navarixin plasma Cmax.
Time Frame: as for outcome 10
Population: Participants with available Cmax data, who complied with the protocol sufficiently to ensure that their data was likely to exhibit the effects of treatment, according to the underlying scientific model. Compliance includes, but is not limited to, exposure to treatment, availability of measurements, and absence of major protocol violations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Navarixin 30 mg + Pembrolizumab 200 mg | Navarixin 100 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 45 | 46
ng/mL | 172 (53.3) | 288 (60.6)

13. Secondary Outcome: Navarixin Trough Plasma Concentration (Ctrough)
Description: Plasma samples from participants with selected advanced/metastatic solid tumors were collected at steady state on Cycle 2 Day 21 to determine navarixin Ctrough. The Arithmetic Mean and CV% are presented.
Time Frame: Cycle 2 Day 21 (Up to approximately 43 days)
Population: Participants with available Ctrough data, who complied with the protocol sufficiently to ensure that their data was likely to exhibit the effects of treatment, according to the underlying scientific model. Compliance includes, but is not limited to, exposure to treatment, availability of measurements, and absence of major protocol violations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Navarixin 30 mg + Pembrolizumab 200 mg | Navarixin 100 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 36 | 35
ng/mL | NA (NA) — Measure Type - Arithmetic Mean: 7.71 Measure of Dispersion - CV%: 10.7% | NA (NA) — Measure Type - Arithmetic Mean: 14.5 Measure of Dispersion - CV%: 77.3%

ADVERSE EVENTS:
Time Frame: All-cause mortality: From randomization up to approximately 27 months; Adverse Events (AEs) from first treatment up to approximately 27 months
Description: All-Cause Mortality was reported for all randomized participants. AEs were reported for all participants who received at least 1 dose of study treatment.
Arm/Group | Navarixin 30 mg + Pembrolizumab 200 mg | Navarixin 100 mg + Pembrolizumab 200 mg
All-Cause Mortality (participants affected / at risk) | 48/52 | 45/55
Serious Adverse Events (participants affected / at risk) | 17/51 | 15/54
Other Adverse Events (participants affected / at risk) | 48/51 | 52/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Navarixin 30 mg + Pembrolizumab 200 mg (N=51) | Navarixin 100 mg + Pembrolizumab 200 mg (N=54)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (7) | 1 (1)
Pseudomonas infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Navarixin 30 mg + Pembrolizumab 200 mg (N=51) | Navarixin 100 mg + Pembrolizumab 200 mg (N=54)
Anaemia (Blood and lymphatic system disorders) | 7 (7) | 5 (6)
Neutropenia (Blood and lymphatic system disorders) | 5 (7) | 9 (12)
Hypothyroidism (Endocrine disorders) | 2 (2) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 9 (10) | 5 (6)
Constipation (Gastrointestinal disorders) | 7 (7) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 7 (7)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (9) | 16 (17)
Vomiting (Gastrointestinal disorders) | 5 (7) | 10 (10)
Asthenia (General disorders) | 5 (7) | 4 (4)
Chills (General disorders) | 1 (1) | 3 (3)
Fatigue (General disorders) | 17 (18) | 14 (14)
Oedema peripheral (General disorders) | 4 (4) | 4 (5)
Pyrexia (General disorders) | 12 (18) | 12 (16)
Pneumonia (Infections and infestations) | 3 (3) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 5 (5)
Urinary tract infection (Infections and infestations) | 5 (9) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 4 (4)
Blood alkaline phosphatase increased (Investigations) | 3 (3) | 4 (4)
Blood creatinine increased (Investigations) | 1 (1) | 3 (3)
Neutrophil count decreased (Investigations) | 7 (11) | 10 (13)
Weight decreased (Investigations) | 6 (6) | 5 (5)
White blood cell count decreased (Investigations) | 3 (3) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 14 (14) | 8 (8)
Dehydration (Metabolism and nutrition disorders) | 4 (5) | 7 (9)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 9 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 10 (11)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Headache (Nervous system disorders) | 8 (8) | 7 (8)
Dysuria (Renal and urinary disorders) | 5 (5) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 8 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (11) | 6 (7)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the sponsor, the investigator agrees to submit all manuscripts or abstracts to the sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/25/NCT03473925/Prot_SAP_000.pdf